CLINICAL TRIAL: NCT07174414
Title: Cilostazol for Prevention of Recurrent Stroke Trial
Acronym: Clarity
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Yale University (Other); University of Cincinnati (Other); Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Maarten Lansberg, Professor of Neurology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 82476; 1UG3NS133209-01A1 (NIH)
Record Dates: First submitted 2025-09-12; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Stroke Recurrence; Myocardial Infarction; Vascular Death; Ischemic Stroke; TIA (Transient Ischemic Attack); Stroke (CVA) or Transient Ischemic Attack; Recurrent Stroke
MeSH Terms: conditions — Myocardial Infarction; Ischemic Stroke; Ischemic Attack, Transient; Stroke | interventions — Cilostazol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masked Statistician and Unmasked statistician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cilostazol 100mg (Experimental): Participants take oral cilostazol until a study endpoint occurs, they reach maximum follow up duration (4 years), the participant withdraws, or the study ends.
  Interventions: Drug: Cilostazol 100 mg
- Placebo (Placebo Comparator): Participants take oral placebo until a study endpoint occurs, they reach maximum follow up duration (4 years), the participant withdraws, or the study ends.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cilostazol 100 mg — Cilostazol 100 mg tablet taken orally twice daily following an initial 2-week period during which cilostazol is dosed at 100 mg tablet taken orally once daily to maximize tolerability.
  Arms: Cilostazol 100mg
Drug: Placebo — Placebo 100 mg tablet twice taken orally daily following an initial 2-week period during which placebo is dosed at 100 mg taken orally once daily to maximize tolerability.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn whether adding cilostazol to aspirin or clopidogrel prevents stroke and heart attack in people who have had a stroke or mini-stroke.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stroke or mini-stroke (also called TIA) within the last 180 days
* Currently taking aspirin or clopidogrel (not both) to prevent another stroke

Exclusion Criteria:

* Had a spontaneous brain bleed within the last 2 years.
* Moderate to severe heart failure.
* Life expectancy is less than 6 months.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2026-08 (Estimated); Primary Completion 2031-07 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular event (MACE) | Up to 4 years after randomization
  Time to stroke (ischemic and hemorrhagic), acute myocardial infarction, or vascular death

SECONDARY OUTCOMES:
Ischemic stroke | Up to 4 years after randomization
  Time to ischemic stroke
Major hemorrhage | Up to 4 years after randomization
  Time to major hemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Lansberg, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnston SC, Easton JD, Farrant M, Barsan W, Conwit RA, Elm JJ, Kim AS, Lindblad AS, Palesch YY; Clinical Research Collaboration, Neurological Emergencies Treatment Trials Network, and the POINT Investigators. Clopidogrel and Aspirin in Acute Ischemic Stroke and High-Risk TIA. N Engl J Med. 2018 Jul 19;379(3):215-225. doi: 10.1056/NEJMoa1800410. Epub 2018 May 16. PMID 29766750
- [Background] Spieler JF, De Pouvourville G, Amarenco P. Cost of a recurrent vs. cost of first-ever stroke over an 18-month period. Eur J Neurol. 2003 Nov;10(6):621-4. doi: 10.1046/j.1468-1331.2003.00665.x. PMID 14641505
- [Background] Engel-Nitz NM, Sander SD, Harley C, Rey GG, Shah H. Costs and outcomes of noncardioembolic ischemic stroke in a managed care population. Vasc Health Risk Manag. 2010 Oct 5;6:905-13. doi: 10.2147/VHRM.S10851. PMID 20957133
- [Background] Serena J, Segura T, Roquer J, Garcia-Gil M, Castillo J; ARTICO Study. The ARTICO study: identification of patients at high risk of vascular recurrence after a first non-cardioembolic stroke. BMC Neurol. 2015 Mar 11;15:28. doi: 10.1186/s12883-015-0278-4. PMID 25884666
- [Background] Nedeltchev K, der Maur TA, Georgiadis D, Arnold M, Caso V, Mattle HP, Schroth G, Remonda L, Sturzenegger M, Fischer U, Baumgartner RW. Ischaemic stroke in young adults: predictors of outcome and recurrence. J Neurol Neurosurg Psychiatry. 2005 Feb;76(2):191-5. doi: 10.1136/jnnp.2004.040543. PMID 15654030
- [Background] Khanevski AN, Bjerkreim AT, Novotny V, Naess H, Thomassen L, Logallo N, Kvistad CE; NOR-STROKE study group. Recurrent ischemic stroke: Incidence, predictors, and impact on mortality. Acta Neurol Scand. 2019 Jul;140(1):3-8. doi: 10.1111/ane.13093. Epub 2019 Apr 11. PMID 30929256
- [Background] Skajaa N, Adelborg K, Horvath-Puho E, Rothman KJ, Henderson VW, Thygesen LC, Sorensen HT. Risks of Stroke Recurrence and Mortality After First and Recurrent Strokes in Denmark: A Nationwide Registry Study. Neurology. 2022 Jan 24;98(4):e329-e342. doi: 10.1212/WNL.0000000000013118. PMID 34845054
- [Background] Oza R, Rundell K, Garcellano M. Recurrent Ischemic Stroke: Strategies for Prevention. Am Fam Physician. 2017 Oct 1;96(7):436-440. PMID 29094912
- [Background] Benjamin EJ, Muntner P, Alonso A, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Das SR, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Jordan LC, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, O'Flaherty M, Pandey A, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Spartano NL, Stokes A, Tirschwell DL, Tsao CW, Turakhia MP, VanWagner LB, Wilkins JT, Wong SS, Virani SS; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2019 Update: A Report From the American Heart Association. Circulation. 2019 Mar 5;139(10):e56-e528. doi: 10.1161/CIR.0000000000000659. No abstract available. PMID 30700139